CLINICAL TRIAL: NCT06699147
Title: Multicenter, Prospective, Observational Study to Evaluate the Post-marketing Efficacy and Safety of Eptq S and Eptq Lidocaine S Applied to the Facial Region
Brief Title: Evaluate the Post-marketing Efficacy and Safety of Eptq S and Eptq Lidocaine S
Status: Completed | Type: Observational
Sponsor: Jetema Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: JT-D-OS-001
Record Dates: First submitted 2024-11-14; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Nasolabial Folds; Mid Face Volume Loss; Lip Volume Enhancement
Keywords: Hyaluronic acid filler; facial region

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Nasolabial Folds: Wrinkle Severity Rating Scale(WSRS) assessed 3 or 4
  Interventions: Device: Hyaluronic Acid (HA)
- Mid-Face Volume: Midface Volume Deficit Scale(MFVDS) assessed 3 or higher
  Interventions: Device: Hyaluronic Acid (HA)
- Lip Volume: Medicis Lip Fullness Scale(MLFS) assessed 1 or 2
  Interventions: Device: Hyaluronic Acid (HA)

INTERVENTIONS:
Device: Hyaluronic Acid (HA) — 6 types of hyaluronic acid(HA) fillers that are differ in HA concentration and lidocaine were used for this study. Each type was applied to different condition or group depending on the investigators medical diagnosis

SUMMARY:
This study in multi-center, prospective and observational study. The purpose of this study is to observe effects and safety of hyaluronic acid filler series, eptq S and eptq Lidocaine S, for facial volume and folds.

DETAILED DESCRIPTION:
Participants for this study are treated with eptq S and eptq Lidocaine S for smoothing nasolabial folds or volumizing mid-face or lips. Treating period is around 24 weeks. Facial volume and wrinkle condition, participants' satisfaction, and safety would be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female adults aged 19 years and older.
* Meet one of the following among individuals who want temporary improvement of facial wrinkles and volume.

  1. Wrinkle Severity Rating Scale score 3 or 4 for Nasolabial fold.
  2. Mid-Face Volume Deficit Scale score 3 or greater.
  3. Medicis Lip Fullness Scale score 1-2. In cases of 2-1) and 2-2), participants must meet both sides (right and left) to be eligible for enrollment.

     For 3), the Medicis Lip Fullness Scale scores 1-2 at the target sites for procedures (upper lip, lower lip, up & down) eligible for enrollment
* Voluntarily agree to participate in this observational study in written consent form.

Exclusion Criteria:

* Received anti-thrombotics (except low-dose aspirin [100 mg, maximum 300 mg/day]) within 2 weeks from screening.
* Currently have or have a history of bleeding disorder.
* applied graft/prosthesis or biomaterials, including hyaluronic acid, polycaprolactone, collagen filler, lifting (threads, laser, etc.), and Botulinum toxin, at the site for indication within 24 weeks from screening.
* Skin disorder or wound infection on the face that affects this study
* Have history of side effects of EMLA cream or equivalent lidocaine agent.
* History of hypersensitivity to hyaluronic acid agent(s).
* Other contraindications as per the [Precautions for Use] in the approved label for the study device.
* Determined as not eligible for the study by the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Beauty Bar Clinics and 8 other clinics in South Korea
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
Nasolabial Folds | 24 weeks
  Percentage(%) of subjects whose Wrinkle Severity Rating Scale was improved during follow-up period compared to the baseline
  (1: No visible fold - 5: Extremly deep fold)
Mid-Face Volume | 24 weeks
  Percentage(%) of subjects whose Mid-face Volume Deficit Scale was improved during follow-up period compared to the base line (0: None - 5: Severe)
Lip Volume | 12 weeks
  Percentage(%) of subjects whose Medicis Lip Fullness Scale was improved during follow-up period compared to the baseline
  (1: Very thin - 5: Very full)

SECONDARY OUTCOMES:
Improvement satisfaction assessment | 24 weeks
  Percentage(%) of subjects whose Global Aesthetic Improvement Scale was improved during follow-up period compared to the base line (-1: Worse - 3: Very much improved)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinics, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No